CLINICAL TRIAL: NCT03004144
Title: Impact of Robotic Assistive Forces on the Performance of Activities of Daily Living
Brief Title: Impact of Assistive Forces on Activities of Daily Living
Acronym: FLOAT-ADL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-01093
Record Dates: First submitted 2016-09-19; First posted 2016-12-28 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2024-11

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- FLOAT-Support (Other)
  Interventions: Other: FLOAT

INTERVENTIONS:
Other: FLOAT

SUMMARY:
This study is a cross-sectional study investigating the impact of assistive forces applied by the body-weight support system "the FLOAT" on the study participants. The study is conducted at the University Hospital Balgrist in Zurich over a period of around 3 years. During this time measurements on approximately 140 able bodied subjects and 60 patients with an incomplete spinal cord injury will take place. The study participants are invited for a single visit of around 140 min duration to the University Hospital Balgrist. During this visit the study participants will repeatedly perform various activities of daily living (free walking, standing up and sitting down, stair climbing and balancing) with and without assistive forces from the body-weight support system. While performing the tasks, the study participants' motions and muscle activities will be measured to evaluate the naturalness of their movements. In addition, the collected data permits us to compare different movement patterns and make conclusions about effective and optimal movement support. Obtaining this knowledge will help us to shape the therapy of these activities to be tailored to the patients and to train these movements with the help of the FLOAT under optimal conditions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with incomplete spinal cord injury (AIS C-D) or able bodied persons
* informed consent as documented by signature
* bodyweight < 120 kg

Exclusion Criteria:

* a significant psychiatric or orthopedic diagnose
* any secondary neurological complications that may impact the outcome variables
* dermatological conditions (pressure ulcers, etc.)
* pacemaker or other implanted, electronic devices
* contraindications for FLOAT training
* inability or unwillingness to provide written informed consent or follow study procedures e.g. due to language problems
* psychological disorders, dementia, etc.
* known or suspected non-compliance, drug or alcohol abuse
* enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-10; Primary Completion 2019-10-24 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
3-dimensional kinematic analyses resulting in a detailed movement profile for each of the performed tasks | Once (single visit) around 140 minutes duration

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik Balgrist, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No